CLINICAL TRIAL: NCT02810340
Title: A Phase 1, Double Blind, Randomized, Controlled Study to Evaluate the Safety and Immunogenicity of a New Meningococcal Conjugate Vaccine Containing Serogroups A,C,Y,W and X in Healthy Adults
Brief Title: Study of Meninigococcal Conjugate Vaccine Containing Serogroups A,C,Y,W and X (MCV5) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAC-046
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Results first posted 2021-03-30 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2019-08

CONDITIONS: Meningococcal Vaccines
MeSH Terms: interventions — Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- MCV-5 with adjuvant (Experimental): Received a single intramuscular injection of Adjuvanted MCV-5.
  Interventions: Biological: Adjuvanted MCV-5
- MCV-5 without adjuvant (Experimental): Received a single intramuscular injection of Non-Adjuvanted MCV-5.
  Interventions: Biological: Non-Adjuvanted MCV-5
- Menactra® (Active Comparator): Received a single intramuscular injection of Menactra.
  Interventions: Biological: Menactra®

INTERVENTIONS:
Biological: Adjuvanted MCV-5 — Contains 5 μg each of N. meningitidis A, C, Y, W, and X polysaccharides, 2.42 mg sucrose, 0.40 mg sodium citrate, 0.098 mg tris (trometamol), 7.8 to 33.4 μg tetanus toxoid, 11.7 to 50.1 μg cross reactive material of diphtheria toxin (CRM), and 125 μg Al3+adjuvant.
  Arms: MCV-5 with adjuvant
Biological: Non-Adjuvanted MCV-5 — Contains 5 μg each of N. meningitidis A, C, Y, W, and X polysaccharides, 2.42 mg sucrose, 0.40 mg sodium citrate, 0.098 mg tris (trometamol), 7.8 to 33.4 μg tetanus toxoid, and 11.7 to 50.1 μg cross reactive material of diphtheria toxin (CRM).
  Arms: MCV-5 without adjuvant
Biological: Menactra® — Menactra® vaccine was a clear to slightly turbid solution supplied in a 0.5 mL single dose vial. Each 0.5 mL dose of vaccine was formulated in sodium phosphate buffered isotonic sodium chloride solution to contain four mcg each of meningococcal A, C, Y, and W-135 polysaccharides conjugated to approximately 48 μg of diphtheria toxoid protein carrier and residual amounts of formaldehyde of less than 2.66 μg (0.000532%), by calculation.
  Arms: Menactra®

SUMMARY:
The primary objective of this study is to evaluate the safety of adjuvanted and non-adjuvanted formulations of MCV-5 vaccine. The secondary objective is to assess the immune response of adjuvanted and non-adjuvanted formulations of MCV-5 vaccine.

DETAILED DESCRIPTION:
Prior to the study, there was no vaccine available against serogroup X of N. meningitidis. This bacterium has caused many outbreaks in Africa and Europe in recent past. It has been responsible for outbreaks between 2006 and 2010 in Kenya, Niger, Togo, Uganda, and Burkina Faso, the latter with at least 1,300 cases of serogroup X meningitis among the 6,732 reported annual cases. The WHO has expressed concerns over the lack of a serogroup X vaccine and has encouraged more research into it. As a result, Serum Institute of India Private Limited (SIIPL) has developed the candidate vaccine MCV-5 (currently renamed NmCV-5), which is a polyvalent conjugate vaccine composed of serogroups A, C, Y, W, and X of Neisseria meningitidis capsular polysaccharides, conjugated to protein carriers, CRM and tetanus toxoid, with aluminum phosphate as an adjuvant. It is intended for the prevention of meningitis and/or septicemia caused by serogroups A, C, Y, W, and X of N. meningitidis in countries where the disease is endemic and causes large epidemics, such as the countries in the African meningitis belt.

The three-group design of the study will allow safety evaluation of the adjuvanted and nonadjuvanted MCV-5 formulations. Menactra® has been chosen as the control vaccine, because of the large safety database accumulated since the vaccine has been introduced in the USA in 2005 and progressively in other countries

ELIGIBILITY:
Inclusion Criteria:

* age 18-45 years
* Written informed consent of volunteers
* Healthy as established by medical history, laboratory evaluation and screening evaluations
* Participants are able to understand and comply with planned study procedures and be available for all study visits
* Female subjects must be of non-childbearing potential (defined as surgically sterile or postmenopausal for more than 1 year), or if of childbearing potential must be practicing abstinence or using an effective licensed method of birth control

Exclusion Criteria:

* Previous vaccination against Neisseria meningitidis.
* Known exposure to Neisseria meningitidis in the past.
* History of meningitis or seizures or any neurological or psychiatric disorder.
* Administration of any other vaccine within 30 days prior or after administration of study vaccines.
* Use of any investigational or non-registered drug or vaccine within 30 days prior to the administration of study vaccines or planned during the study.
* History of allergic disease or known hypersensitivity to any component of the three study vaccines.
* History of Serious Adverse Reactions following administration of Tetanus Toxoid, Diphtheria Toxoid or CRM containing vaccines.
* History of Guillan-Barré syndrome.
* Confirmed or suspected immunosuppressive or immune-deficient condition. 10. A family history of congenital or hereditary immunodeficiency.
* Chronic administration (defined as more than 14 days) of immune-suppressants or other immune-modifying agents within six months prior to administration of study vaccine.
* 12. Laboratory confirmed infection of either hepatitis B virus (HBs Ag positive on ELISA), hepatitis C virus (anti-HCV positive on ELISA as well as PCR) or human immunodeficiency virus (HIV on ELISA).
* Major congenital defects or serious chronic illness.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by medical history, physical examination or laboratory screening tests.
* Known bleeding disorders.
* Administration of immunoglobulins and/or any blood products within the three months preceding the administration of study vaccines or planned administration during the vaccine period.
* History (within the past year) or signs of alcohol or substance abuse.
* Pregnancy or lactation.
* A Body Mass Index (BMI) equal to or above 30.
* Any other condition, which in the opinion of the investigator, might interfere with the study objectives, jeopardize the safety or rights of the participant or making it unlikely the participant could complete the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-10-13 (Actual); Study Completion 2017-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilbur Chen, MD,MS, Principal Investigator — University of Maryland Scool of Medicine, Baltimore
Locations (1):
- Center for Vaccine Development, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Chen WH, Neuzil KM, Boyce CR, Pasetti MF, Reymann MK, Martellet L, Hosken N, LaForce FM, Dhere RM, Pisal SS, Chaudhari A, Kulkarni PS, Borrow R, Findlow H, Brown V, McDonough ML, Dally L, Alderson MR. Safety and immunogenicity of a pentavalent meningococcal conjugate vaccine containing serogroups A, C, Y, W, and X in healthy adults: a phase 1, single-centre, double-blind, randomised, controlled study. Lancet Infect Dis. 2018 Oct;18(10):1088-1096. doi: 10.1016/S1473-3099(18)30400-6. Epub 2018 Aug 14. PMID 30120069

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MCV-5 With Adjuvant | MCV-5 Without Adjuvant | Menactra®
Started | 20 | 20 | 20
Completed | 19 | 19 | 19
Not Completed | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Incarceration | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MCV-5 With Adjuvant | MCV-5 Without Adjuvant | Menactra® | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (6.38) | 30.4 (7.23) | 33.1 (7.43) | 32.5 (7.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 6 | 23
  Male | 12 | 11 | 14 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 20 | 19 | 20 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 9 | 13 | 33
  White | 5 | 10 | 6 | 21
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: inches] | 67.2 (2.90) | 66.8 (2.88) | 68.6 (4.18) | 67.5 (3.41)
Weight [Mean (Standard Deviation); unit: pounds] | 158.2 (24.56) | 150.0 (26.87) | 174.6 (27.58) | 160.9 (27.90)

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants Experiencing Solicited Events
Description: Solicited reactions (reactogenicity) were collected following vaccination through Day 7. If a solicited sign or symptom had started during the seven days post-vaccination period and continued beyond Day 7, it was still assessed as a solicited reaction.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | MCV-5 With Adjuvant | MCV-5 Without Adjuvant | Menactra®
Number analyzed (Participants) | 20 | 20 | 20
Participants
  Solicited AE: Pain at injection site | 12 | 10 | 7
  Solicited AE: Erythema at injection site | 0 | 1 | 1
  Solicited AE: Swelling at injection site | 1 | 1 | 1
  Solicited AE: Any local symptom | 12 | 10 | 8
  Solicited AE: Fever | 0 | 0 | 0
  Solicited AE: Headache | 5 | 3 | 3
  Solicited AE: Fatigue/malaise | 3 | 3 | 2
  Solicited AE: Joint pain/arthralgia | 1 | 1 | 2
  Solicited AE: Muscle pain/myalgia | 2 | 6 | 3
  Solicited AE: Diarrhea | 3 | 1 | 2
  Solicited AE: Anorexia | 1 | 0 | 1
  Solicited AE: Chills | 1 | 1 | 1
  Solicited AE: Vomiting | 0 | 1 | 1
  Solicited AE: Any systemic symptom | 8 | 8 | 8
  Solicited AE: Any systemic or local symptom | 13 | 12 | 10

2. Primary Outcome: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events, by Severity
Description: Adverse events (AE) were collected through day 28. Safety clinical laboratory evaluations were performed at Screening and at Day 8 and included: hemoglobin (HgB), white blood cells (WBC), platelet counts, alanine transaminase (ALT), albumin, total bilirubin, and creatinine. In addition, screening laboratory tests included serum HCG pregnancy tests for females of childbearing potential only, and screening for human immunodeficiency virus (HIV), hepatitis C virus (HCV), and hepatitis B virus (HBV) infection. AE severity was graded as per the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0, November 2014, of the US National Institute of Health.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | MCV-5 With Adjuvant | MCV-5 Without Adjuvant | Menactra®
Number analyzed (Participants) | 20 | 20 | 20
Participants
  Mild | 1 | 2 | 5
  Moderate | 2 | 1 | 2
  Severe | 0 | 1 | 0

3. Primary Outcome: Number of Subjects Experiencing Serious Adverse Events
Description: Serious adverse events (AE) were collected 6 months post-immunization. Safety clinical laboratory evaluations were performed at Screening and at Day 8 and included: hemoglobin (HgB), white blood cells (WBC), platelet counts, alanine transaminase (ALT), albumin, total bilirubin, and creatinine. In addition, screening laboratory tests included serum HCG pregnancy tests for females of childbearing potential only, and screening for human immunodeficiency virus (HIV), hepatitis C virus (HCV), and hepatitis B virus (HBV) infection.
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | MCV-5 With Adjuvant | MCV-5 Without Adjuvant | Menactra®
Number analyzed (Participants) | 20 | 20 | 20
Participants | 0 | 0 | 0

4. Secondary Outcome: Number and Percentage of Participants With Seroconversion for Meningococcal Polysaccharide A, C, Y, W and X Specific Antibodies
Description: Defined as a ≥4-fold increase in post-immunization rabbit complement serum bactericidal activity (rSBA) titer between baseline and 28 days post-vaccination. The rSBA assay (previously validated for serogroups A, C, Y, and W) was performed at the Vaccine Evaluation Unit at Public Health England (PHE) in Manchester, United Kingdom.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | MCV-5 With Adjuvant | MCV-5 Without Adjuvant | Menactra®
Number analyzed (Participants) | 20 | 20 | 20
Participants
  Meningococcal Polysaccharide A | 17 | 14 | 16
  Meningococcal Polysaccharide C | 19 | 20 | 17
  Meningococcal Polysaccharide Y | 19 | 19 | 15
  Meningococcal Polysaccharide W | 20 | 19 | 16
  Meningococcal Polysaccharide X | 19 | 17 | 1

5. Secondary Outcome: Number and Percentage of Participants With Seroprotection for Meningococcal Polysaccharide A, C, Y, W and X (Antibody Titer ≥1:8), at Baseline and After 28 Days
Description: Seroprotection defined as a titer ≥1:8 in post-immunization rabbit complement serum bactericidal activity (rSBA) titer between baseline and 28 days post-vaccination. The rSBA assay (previously validated for serogroups A, C, Y, and W) was performed at the Vaccine Evaluation Unit at Public Health England (PHE) in Manchester, United Kingdom.
Time Frame: Baseline and Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | MCV-5 With Adjuvant | MCV-5 Without Adjuvant | Menactra®
Number analyzed (Participants) | 20 | 20 | 20
Participants
  Meningococcal Polysaccharide A: Baseline | 15 | 17 | 10
  Meningococcal Polysaccharide A: Day 29 | 20 | 20 | 20
  Meningococcal Polysaccharide C: Baseline | 9 | 3 | 4
  Meningococcal Polysaccharide C: Day 29 | 20 | 20 | 18
  Meningococcal Polysaccharide Y: Baseline | 6 | 9 | 12
  Meningococcal Polysaccharide Y: Day 29 | 19 | 20 | 20
  Meningococcal Polysaccharide W: Baseline | 5 | 9 | 8
  Meningococcal Polysaccharide W: Day 29 | 20 | 20 | 18
  Meningococcal Polysaccharide X: Baseline | 5 | 3 | 2
  Meningococcal Polysaccharide X: Day 29 | 19 | 20 | 2

6. Secondary Outcome: Number and Percentage of Participants With Seroprotection for Meningococcal Polysaccharide A, C, Y, W and X (Antibody Titer ≥1:128), at Baseline and After 28 Days
Description: Seroprotection defined as a titer ≥1:128 in post-immunization rabbit complement serum bactericidal activity (rSBA) titer between baseline and 28 days post-vaccination. The rSBA assay (previously validated for serogroups A, C, Y, and W) was performed at the Vaccine Evaluation Unit at Public Health England (PHE) in Manchester, United Kingdom.
Time Frame: Baseline and Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | MCV-5 With Adjuvant | MCV-5 Without Adjuvant | Menactra®
Number analyzed (Participants) | 20 | 20 | 20
Participants
  Meningococcal Polysaccharide A: Baseline | 15 | 17 | 10
  Meningococcal Polysaccharide A: Day 29 | 20 | 20 | 20
  Meningococcal Polysaccharide C: Baseline | 5 | 2 | 4
  Meningococcal Polysaccharide C: Day 29 | 19 | 20 | 17
  Meningococcal Polysaccharide Y: Baseline | 6 | 9 | 12
  Meningococcal Polysaccharide Y: Day 29 | 19 | 20 | 20
  Meningococcal Polysaccharide W: Baseline | 5 | 9 | 7
  Meningococcal Polysaccharide W: Day 29 | 20 | 20 | 18
  Meningococcal Polysaccharide X: Baseline | 3 | 3 | 2
  Meningococcal Polysaccharide X: Day 29 | 19 | 20 | 2

7. Secondary Outcome: Geometric Mean Titer (GMT) of Meningococcal Polysaccharide A, C, Y, W and X Specific Antibodies at Baseline and After 28 Days
Description: Measured with rabbit complement serum bactericidal activity (rSBA) assay at baseline and 28 days post-vaccination. The rSBA assay (previously validated for serogroups A, C, Y, and W) was performed at the Vaccine Evaluation Unit at Public Health England (PHE) in Manchester, United Kingdom.
Time Frame: Baseline and Day 29
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | MCV-5 With Adjuvant | MCV-5 Without Adjuvant | Menactra®
Number analyzed (Participants) | 20 | 20 | 20
titer
  Meningococcal Polysaccharide A: Baseline | 187 [49.6 to 708] | 350 [119 to 1025] | 33.1 [8.42 to 130]
  Meningococcal Polysaccharide A: Day 29 | 6889 [3767 to 12596] | 5595 [3324 to 9418] | 3214 [1978 to 5222]
  Meningococcal Polysaccharide C: Baseline | 9.85 [3.77 to 25.7] | 4.29 [2.01 to 9.15] | 5.66 [2.15 to 14.9]
  Meningococcal Polysaccharide C: Day 29 | 4096 [1720 to 9756] | 6208 [3579 to 10771] | 388 [139 to 1085]
  Meningococcal Polysaccharide Y: Baseline | 10.2 [3.03 to 34.4] | 24.3 [6.16 to 95.4] | 53.8 [14.2 to 204]
  Meningococcal Polysaccharide Y: Day 29 | 4545 [1700 to 12149] | 9410 [4935 to 17942] | 2353 [1302 to 4251]
  Meningococcal Polysaccharide W: Baseline | 8.00 [2.44 to 26.2] | 26.9 [6.19 to 117] | 13.9 [4.16 to 46.6]
  Meningococcal Polysaccharide W: Day 29 | 8192 [3439 to 19513] | 11191 [6720 to 18635] | 1261 [388 to 4091]
  Meningococcal Polysaccharide X: Baseline | 6.28 [2.44 to 16.1] | 5.28 [1.89 to 14.8] | 3.36 [1.76 to 6.43]
  Meningococcal Polysaccharide X: Day 29 | 1351 [577 to 3165] | 1607 [892 to 2895] | 3.14 [1.73 to 5.71]

8. Secondary Outcome: Geometric Mean Fold Change in Meningococcal Polysaccharide A, C, Y, W and X Specific Antibody Titers
Description: as for outcome 7
Time Frame: 28 days
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | MCV-5 With Adjuvant | MCV-5 Without Adjuvant | Menactra®
Number analyzed (Participants) | 20 | 20 | 20
fold change
  Meningococcal Polysaccharide A | 36.8 [9.97 to 135] | 16.0 [5.74 to 44.6] | 97.0 [22.7 to 414]
  Meningococcal Polysaccharide C | 416 [125 to 1381] | 1448 [507 to 4138] | 68.6 [20.2 to 233]
  Meningococcal Polysaccharide Y | 446 [127 to 1560] | 388 [77.7 to 1937] | 43.7 [11.7 to 164]
  Meningococcal Polysaccharide W | 1024 [359 to 2918] | 416 [94.5 to 1829] | 90.5 [20.7 to 396]
  Meningococcal Polysaccharide X | 215 [66.1 to 701] | 304 [90.1 to 1029] | 0.93 [0.49 to 1.78]

ADVERSE EVENTS:
Time Frame: 7 days for solicited adverse events; 28 days for unsolicited non-serious adverse events; 180 days for serious adverse events.
Description: No deaths and no serious adverse events were reported in this study. The Other Adverse Events table includes only unsolicited adverse events reporting because per study statistical analysis plan, unsolicited adverse events and solicited adverse events were presented separately. For a complete count of the solicited events, please refer to primary outcome safety tables.
Arm/Group | MCV-5 With Adjuvant | MCV-5 Without Adjuvant | Menactra®
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 14/20 | 13/20 | 11/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MCV-5 With Adjuvant (N=20) | MCV-5 Without Adjuvant (N=20) | Menactra® (N=20)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (3) | 3 (3) | 2 (2)
Injection site discolouration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 1 (1)
Injection site pain (General disorders) | 12 (12) | 10 (10) | 7 (7)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 1 (1) | 1 (1) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) | 3 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/40/NCT02810340/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT02810340/SAP_001.pdf